CLINICAL TRIAL: NCT04635202
Title: Effect of Elliptical Training on Lipids, Glucose and Insulin Homeostasis in Metabolic Syndrome
Brief Title: Effect of Elliptical Training on Metabolic Homeostasis in Metabolic Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ali Mohamed Ali ismail, lecturer of Physical Therapy for Cardiovascular / Respiratory Disorder and Geriatrics, Faculty of Physical Therapy, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/002896
Record Dates: First submitted 2020-11-13; First posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Experimental): patients (n=30) in this group will receive 16 weeks of elliptical training on elliptical trainer, 3 times per week. the training will start with 5 minutes warming up at 50 % of maximal heart rate (MHR), 20-minute continuous ET at 70% of MHR, 12 minutes (4×3) intervals at 90% of MHR with a 3-minute active recovery at 70% of MHR between intervals, and finally 5-minute cool-down period at 50% of MHR
  Interventions: Behavioral: exercise training on elliptical device
- Group B (control group) (Other): patients (n=30) in this group will receive general advises on maintaining physical activities
  Interventions: Behavioral: group B (control group)

INTERVENTIONS:
Behavioral: exercise training on elliptical device — This group (n=30) will receive aerobic training on an elliptical trainer for 16 weeks (3 sessions per week). The session will start with 5 minutes warming up at 50 % of maximal heart rate (MHR), 20-minute continuous ET at 70% of MHR, 12 minutes (4×3) intervals at 90% of MHR with a 3-minute active recovery at 70% of MHR between intervals, and finally 5-minute cool-down period at 50% of MHR
  Other Names: group A
  Arms: group A
Behavioral: group B (control group) — this group will receive general advises on maintaining physical activities for 16 weeks without any additional supervised training
  Arms: Group B (control group)

SUMMARY:
The growing prevalence of metabolic syndrome (MetS) in the worldwide is becoming a serious health problem and economic burden. MetS has become a crucial risk factor for the development of type 2 diabetes mellitus (T2DM) and cardiovascular diseases (CVD). The rising rates of CVD and diabetes, which are the two leading causes of death. To prevent the progression of MetS to diabetes and CVD, regular physical activity is required.

Elliptical trainer device is a relatively new modality of exercise and is advertised to be superior to a treadmill because of the low joint impact and the more reasonable costs of an elliptical trainer compared to a treadmill. Additional quantitative research is needed to further evaluate the effectiveness of elliptical trainers and the physiological and perceptual responses to the machine.

DETAILED DESCRIPTION:
Forty sedentary MeTS patients (from both sexes) will be randomly divided to group A and group B.

-Group A (Elliptical training group): This group (n=20) will receive aerobic training on an elliptical trainer for 16 weeks (3 sessions per week). The session will start with 5 minutes warming up at 50 % of maximal heart rate (MHR), 20-minute continuous ET at 70% of MHR, 12 minutes (4×3) intervals at 90% of MHR with a 3-minute active recovery at 70% of MHR between intervals, and finally 5-minute cool-down period at 50% of MHR.

Group B: this group will continue their normal daily physical activities without any additional training

ELIGIBILITY:
Inclusion Criteria:

* The MeTS subjects who will have three or more of the following criteria: 1) waist circumference more than 102 cm, triglycerides more than 150 mg/dL, 3) blood pressure (BP) more than 130/85 mmHg, 4) high-density lipoprotein (HDL) less than 40 mg/dL, .

Exclusion criteria:

* Renal, pulmonary, cardiac, vascular, respiratory, hepatic, autoimmune disorders.
* Smoker, addictive, cancer, and alcoholic patients.
* Lower limb arthritis or any orthopaedic problem will hinder the training.
* Participation in any type of sport training in the previous 6 months.
* Pregnant or lactating women.
* Patients with thyroid gland dysfunction.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — self-representation of gender identity.
Enrollment: 60 (Estimated)
Dates: Start 2020-09-09 (Actual); Primary Completion 2021-05-15 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Triglycerides | It will be measured after 16 weeks of training
  Triglycerides is one of lipid profile indicators
high density lipoprotein | It will be measured after 16 weeks of training
  high density lipoprotein is one of lipid profile indicators

SECONDARY OUTCOMES:
Systolic blood pressure | It will be measured after 16 weeks of training
  It will be measured via Sphygmomanometer
diastolic blood pressure | It will be measured after 16 weeks of training
  It will be measured via Sphygmomanometer
Fasting blood glucose | It will be measured after 16 weeks of training
  It will be measured via a blood glucose meter
Insulin | It will be measured after 16 weeks of training
  it will be measured via a blood sample
The HOMA-IR (Homeostatic Model Assessment for Insulin Resistance | It will be measured after 16 weeks of training
  HOMA-IR = [fasting insulin (μU/mL)
  × fasting glucose (mmol)]/22.5
Waist circumference | It will be measured after 16 weeks of training
  it will be measured by inelastic tape at the umbilicus level
weight | It will be measured after 16 weeks of training
  the weight scale will be used
Leg strength test | It will be measured after 16 weeks of training
  will be assessd by leg dynamometer
% body fat | It will be measured after 16 weeks of training
  percentage of body fat composition

CONTACTS AND LOCATIONS:
Overall Officials: Ali Ismail, lecturer, Principal Investigator — Cairo University
Locations (1):
- Faculty of Physical Therapy Cairo University, Giza, Dokki, Egypt